CLINICAL TRIAL: NCT06310135
Title: Filtered Eyewear to Prevent Light-induced Melatonin Suppression While Maintaining Visual Performance and Alertness in Night-shift Working Nurses - Aim 1
Brief Title: Filtered Eyewear to Prevent Light-induced Melatonin Suppression - Aim 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-23-00816
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Unfiltered Monocular (Experimental): Unfiltered monocular with the non-dominant eye occluded.
  Interventions: Device: Unfiltered Eyewear
- Filtered Binocular (Experimental): Filtered binocular with both eyes filtered.
  Interventions: Device: Filtered Eyewear
- Filtered Monocular (Experimental): Filtered monocular with non-dominant eye filtered, the other non-filtered.
  Interventions: Device: Filtered Eyewear
- Unfiltered Binocular (Experimental): Unfiltered binocular - neither eye will be filtered.
  Interventions: Device: Unfiltered Eyewear
- Dim Light Control (Placebo Comparator): Dim light with no filters.
  Interventions: Other: No Filters

INTERVENTIONS:
Device: Filtered Eyewear — Filtered binocular viewing condition will be produced by eyeglasses frames with orange-tinted blue-blocking filter, eliminating all optical radiation for wavelengths shorter than 540 nm. For the filtered monocular condition, only the lens on the eyeglasses frame on the non-dominant eye will be tinted with the blue-blocking filter.
  Arms: Filtered Binocular; Filtered Monocular
Device: Unfiltered Eyewear — For the unfiltered binocular, the subjects will wear transparent eyeglasses frames with no optical power. Unfiltered monocular vision will be produced by an opaque eyepatch occluding the non-dominant eye.
  Arms: Unfiltered Binocular; Unfiltered Monocular
Other: No Filters — Dim lights with no filters.
  Arms: Dim Light Control

SUMMARY:
The aim of this study is to determine the relative effectiveness of monocular and binocular light exposures, with and without selective blue-blocking filtering, on nocturnal melatonin suppression, subjective sleepiness, and visual performance of night shift workers.

DETAILED DESCRIPTION:
Over the course of six, 5-hour study nights, 30 participants will be randomized to 6 study conditions, 1) binocular dim-light control unfiltered, (2) monocular dim-light control (one eye occluded), (3) unfiltered binocular, (4) unfiltered monocular (non-dominant eye occluded), (5) filtered binocular (both eyes filtered), (6) filtered monocular (non-dominant eye filtered, the other non-filtered). Saliva samples will be collected every 30 minutes for melatonin levels. Participants will also be asked to provide subjective sleepiness and visual performance will be assessed. Study nights will be separated by one week and each participant will be randomized to one of the six study conditions each night. All participants will see all conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Bipolar disorder
* Seasonal depression
* Diabetes
* High blood pressure
* History of cancer
* Obstructing cataracts
* Macular degeneration
* Diabetic retinopathy
* Glaucoma
* Use of melatonin supplements
* Use of beta blockers
* Use of sleep medications
* Use of antidepressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Melatonin Levels AUC | Each night for 6 study nights
  Melatonin levels to assess Melatonin Suppression. Saliva samples will be collected every 30 minutes for melatonin levels.

SECONDARY OUTCOMES:
Karolinska Sleepiness scale to measure Subjective Sleepiness | Each night for 6 study nights
  Subjective sleepiness will be measured using the Karolinska Sleepiness scale. This 9-point scale scores range from 1-9, where 1 = "very alert," 3 = "alert," 5 = "neither alert nor sleepy," 7 = "sleepy, but no difficulty remaining awake," and 9 = "very sleepy, fighting sleep, an effort to remain awake." Full scale from 1-9. A higher number indicates greater sleepiness.
Numerical Verification Task (NVT) | Each night for 6 study nights
  The NVT requires participants to compare 2 lists of 20 pairs of 5-digit numerals at 2 contrasts (0.2 and 0.8), and the response time required to complete the task is recorded as the performance measure. A faster response time indicates better visual performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Light and Health Research Center, Menands, New York, United States

IPD SHARING:
Plan to Share IPD: No
overall results will be shared, not individual results